CLINICAL TRIAL: NCT03337204
Title: Enhancing the Health-Promoting Effects of Older Adults' Activity Portfolios: The Development, Feasibility and Initial Efficacy of an Ecologically Sensitive Intervention
Brief Title: The Engaged4Life Study: Enhancing the Health-Promoting Effects of Older Adults' Activity Portfolios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-003; P30AG048785 (NIH)
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engaged4Life (Experimental): Participants randomly assigned to this group receive: 1) technology-assisted self-monitoring of daily activity via a Fitbit Zip worn daily (for 8 weeks) and a daily tablet self-report survey (completed for a 7-day period at baseline and a second 7-day period 4-weeks later); and 2) a one-time, 3hr workshop and peer mentoring (via phone 2X/week for 3 weeks). The workshop includes psychoeducation on the relationship between active engagement and health and well-being and a goal setting activity focused on carefully assessing and then make improvements upon existing "activity portfolios". Peer mentors provide support as participants implement their goals.
  Interventions: Behavioral: Technology-assisted self-monitoring; Behavioral: Workshop and Peer Mentoring
- Technology-assisted self-monitoring only (Active Comparator): Participants randomly assigned to this group receive: 1) technology-assisted self-monitoring of daily activity via a Fitbit Zip worn daily (for 8 weeks) and a daily tablet self-report survey (completed for a 7-day period at baseline and a second 7-day period 4-weeks later). While it is expected that wearing the Fitbit and raising consciousness of activity engagement may initially result in behavior change, it is not expected to have a sustained impact on outcomes over time.
  Interventions: Behavioral: Technology-assisted self-monitoring

INTERVENTIONS:
Behavioral: Technology-assisted self-monitoring — Participants receive a Fitbit Zip, an iPad Mini tablet device, training on how to use the Fitbit and iPad, and are asked to complete brief surveys each night on their activity engagement that day (for two 7-day periods).
Behavioral: Workshop and Peer Mentoring — Participants receive a 3-hour Engaged4Life Workshop (psychoeducation + goal setting) and one-on-one peer mentoring via phone 2X/week for 3 weeks.
  Arms: Engaged4Life

SUMMARY:
This study designs and tests a multi-component intervention- Engaged4Life- designed to enhance physical activity (PA), cognitive activity (CA), social interaction (SI) and personal meaning (PM) in low-engaged community-dwelling older adults' everyday life activities through: 1) technology-assisted self-monitoring of PA, CA, SI, and PM activity engagement, 2) psycho-education + goal setting (via a 3-hour workshop), and 3) one-on-one peer mentoring (via phone 2X/week for 3 weeks) to support goal implementation. 15 adults age 65 or older will be randomized to receive all 3 intervention components and 15 to receive only the technology-assisted self-monitoring component.

DETAILED DESCRIPTION:
The Social Model of Health Promotion posits that physical, cognitive, and social activity embedded within activities can help maintain or even restore cognitive and functional health in later life and stimulating activities that carry personal meaning or confer a sense of purpose may have stronger health-promoting effects than activities that are just stimulating. While the Experience Corps program-a community volunteering program for older adults designed to explicitly embed these characteristics-is an effective model for health-promotion, this program is not, as of yet, widely accessible. Further, formal volunteering is not always an activity that is attractive or accessible for older adults, and other interventions aimed at promoting social role involvement among older adults have shown only limited effectiveness in doing so. Thus, the current study explores whether it is possible to create an individually-tailored intervention that encourages older adults to 1) carefully examine their existing "activity portfolios" (technology-assisted self-monitoring), 2) empowers them with the knowledge and skills to make improvements upon their "activity portfolios" by enhancing/supplementing activities in ways that increase their overall levels of physical activity, cognitive activity, social interaction, and personal meaning (psycho-education + goal setting via a workshop), and 3) provides social support through peers in implementing their goals (one-on-one peer mentoring). Targeting a sample of community dwelling older adults who are at-risk for adverse cognitive and physical health outcomes due to their sedentary activity levels, we aim to influence positive changes in overall health and well-being in a way that is more practical, effective, and sustainable than prior interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 or older
* Low-to-moderate engagement levels as determined by a score of <10 on a modified version of the Health Enhancement Lifestyle Profile (HELP) (Hwang, 2010), where only the domains of exercise, social and productive activity, and leisure were included
* A resident of Waltham, MA
* Willing to be randomly assigned to study arm
* Available for relevant study dates

Exclusion Criteria:

* Age of 64 or younger
* Living in an assisted living or nursing home facility
* Significant cognitive impairment (those with >2 errors on the six-item screener by Callahan, Unverzagt, Hui, Perkins, & Hendrie, 2002)
* Reports that a doctor has told them that it is unsafe to participate in physical activity

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2015-11-03 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
Physical Activity: Steps per day | worn daily for 8 weeks
  Measured using the Fitbit Zip pedometer

SECONDARY OUTCOMES:
Cognitive activity (CA)(assessed daily) | asked daily for 7 days at baseline and again for 7 days during week 4
  Cognitive activity (CA) assessed daily was measured as respondents' assessment of the number of cognitively stimulating activities they had participated in that day from a list of 13 activities plus one possible write-in "other" activity.
Social interaction (SI) (assessed daily) | asked daily for 7 days at baseline and again for 7 days during week 4
  Social interaction (SI) questions focused on the quantity (the number of social interactions the respondent had that day, including in-person, by telephone, or by video, but NOT including email, text, or social media) and the quality (whether the participant had a problematic social interaction that day and the perceived stress of the problematic social interaction; and whether the participant had a positive social interaction that day and the perceived positivity of that social interaction) of daily social interactions.
Personal meaning (PM) (assessed daily) | asked daily for 7 days at baseline and again for 7 days during week 4
  Respondents were asked 4 questions around whether they did anything that day that 1) benefited others, 2) left them feeling personally satisfied or accomplished, 3) felt significant in the broader scheme of things, or 4) was personally meaningful. Response options included 0 (not at all), 1 (to some extent), and 3 (to a great extent). Respondents were also asked a more global question: How much did you feel your life had purpose today? Th response scale ranged from 1 to 7 .

CONTACTS AND LOCATIONS:
Overall Officials: Christina J Costa, PhD, Principal Investigator — Boston College

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Callahan CM, Unverzagt FW, Hui SL, Perkins AJ, Hendrie HC. Six-item screener to identify cognitive impairment among potential subjects for clinical research. Med Care. 2002 Sep;40(9):771-81. doi: 10.1097/00005650-200209000-00007. PMID 12218768
- [Background] Hwang JE. Promoting healthy lifestyles with aging: development and validation of the Health Enhancement Lifestyle Profile (HELP) using the Rasch measurement model. Am J Occup Ther. 2010 Sep-Oct;64(5):786-95. doi: 10.5014/ajot.2010.09088. PMID 21073109
- [Background] Heaven B, Brown LJ, White M, Errington L, Mathers JC, Moffatt S. Supporting well-being in retirement through meaningful social roles: systematic review of intervention studies. Milbank Q. 2013 Jun;91(2):222-87. doi: 10.1111/milq.12013. PMID 23758511
- [Background] Fried LP, Carlson MC, Freedman M, Frick KD, Glass TA, Hill J, McGill S, Rebok GW, Seeman T, Tielsch J, Wasik BA, Zeger S. A social model for health promotion for an aging population: initial evidence on the Experience Corps model. J Urban Health. 2004 Mar;81(1):64-78. doi: 10.1093/jurban/jth094. PMID 15047786
- [Background] Fried LP, Carlson MC, McGill S, Seeman T, Xue QL, Frick K, Tan E, Tanner EK, Barron J, Frangakis C, Piferi R, Martinez I, Gruenewald T, Martin BK, Berry-Vaughn L, Stewart J, Dickersin K, Willging PR, Rebok GW. Experience Corps: a dual trial to promote the health of older adults and children's academic success. Contemp Clin Trials. 2013 Sep;36(1):1-13. doi: 10.1016/j.cct.2013.05.003. Epub 2013 May 13. PMID 23680986
- [Background] Jenkinson CE, Dickens AP, Jones K, Thompson-Coon J, Taylor RS, Rogers M, Bambra CL, Lang I, Richards SH. Is volunteering a public health intervention? A systematic review and meta-analysis of the health and survival of volunteers. BMC Public Health. 2013 Aug 23;13:773. doi: 10.1186/1471-2458-13-773. PMID 23968220